CLINICAL TRIAL: NCT01935492
Title: 8 Continuous vs 8 Intermittent Cycles in First and Second Line Treatment of Patients With HER2/Neu Negative, Incurable, Metastatic or Unresectable Locally Advanced Breast Cancer.
Brief Title: 8 Continuous vs 8 Intermittent Cycles in First and Second Line in HER2/Neu Neg Metastatic Breast Cancer
Acronym: Stop&Go
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Roche Pharma AG (Industry); Teva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2010-02 Stop&Go study; NTR2589 (Registry Identifier: Nederlands Trialregister)
Record Dates: First submitted 2010-11-26; First posted 2013-09-05 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Metastatic Breast Cancer
Keywords: metastatic breast cancer; HER2/neu negative; paclitaxel; bevacizumab; liposomal doxorubicine; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Bevacizumab; liposomal doxorubicin; Capecitabine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8 cycles of Paclitaxel & bevacizumab (Active Comparator): 8 cycles of Paclitaxel: 90 mg/m2 IV on days 1, 8 and 15 every 28 days & Bevacizumab: 10 mg/kg IV on days 1 and 15 every 28 days
  Interventions: Drug: Paclitaxel, Bevacizumab, liposomal doxorubicin, Capecitabine
- 2 x 4 cycles of Paclitaxel & bevacizumab (Active Comparator): intermittent 2x4 cycles of Paclitaxel: 90 mg/m2 IV on days 1, 8 and 15 every 28 days & Bevacizumab: 10 mg/kg IV on days 1 and 15 every 28 days
  Interventions: Drug: Paclitaxel, Bevacizumab, liposomal doxorubicin, Capecitabine

INTERVENTIONS:
Drug: Paclitaxel, Bevacizumab, liposomal doxorubicin, Capecitabine — 1. st line:
     * Paclitaxel and bevacizumab: 8 cycles, unless PD or unacceptable toxicity occurs earlier.
     * Bevacizumab until PD or unacceptable toxicity
     * At PD patients will go to the 2nd treatment line.
  2. nd line:
     * Non-pegylated liposomal doxorubicin (Myocet®) (or capecitabine): 8 cycles, unless PD or unacceptable toxicity occurs earlier.
     * At PD patients will go to the 3rd treatment line. If possible, it is advised to cross-over from 2nd line non-pegylated liposomal doxorubicin to 3rd line capecitabine.
  Other Names: Non-pegylated liposomal doxorubicin (Myocet®)
  Arms: 8 cycles of Paclitaxel & bevacizumab
Drug: Paclitaxel, Bevacizumab, liposomal doxorubicin, Capecitabine — Arm B
  1. st line
     * Paclitaxel and bevacizumab: 4 cycles, unless PD or unacceptable toxicity
     * Bevacizumab until PD or unacceptable toxicity
     * At PD < 3 months after last paclitaxel start 2nd treatment line.
     * At PD ≥ 3 months after last paclitaxel, start another 4 cycles
     * Bevacizumab until the next PD or unacceptable toxicity
     * At the next PD start the 2nd treatment line.
  2. nd line:
     * Myocet® or capecitabine: 4 cycles, unless PD or unacceptable toxicity
     * At PD < 3 months start the 3rd treatment line. If possible, advised to cross-over from 2nd line Myocet® to 3rd line capecitabine.
     * At PD ≥ 3 months after last administration of Myocet® or capecitabine, start another 4 cycles of Myocet® or capecitabine
     * At the next PD start 3rd treatment line.
  Other Names: Non-pegylated liposomal doxorubicin (Myocet®):
  Arms: 2 x 4 cycles of Paclitaxel & bevacizumab

SUMMARY:
An open randomized phase III study to compare 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy in first line treatment, in combination with bevacizumab, and second line treatment of patients with HER2/neu negative, incurable, metastatic or unresectable locally advanced breast cancer.

DETAILED DESCRIPTION:
The primary goal of this non-inferiority trial is to determine if the results obtained with a intermittent chemotherapy regimen (2 x 4 cycles of paclitaxel) are not inferior to the results of a continuous chemotherapy regimen (8 cycles of paclitaxel), both combined with bevacizumab in first line treatment of patients with HER2/neu negative, incurable, metastatic or unresectable locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years old.
* Patients with HER2/neu negative, incurable, metastatic or unresectable locally advanced breast cancer, who are candidates for chemotherapy.
* Patients with measurable or evaluable-only (RECIST 1.1)
* Documented Estrogen Receptor (ER) / Progesteron Receptor (PR) status.
* HER2/neu-negative disease
* Patients with an ECOG Performance Status ≤ 2.
* Life expectancy of > 12 weeks.
* Signature of Informed Consent Form

Exclusion Criteria:

* Previous chemotherapy for HER2/neu negative, incurable, metastatic or unresectable locally advanced breast cancer.
* Prior hormonal therapy for HER2/neu negative, incurable, metastatic or unresectable locally advanced breast cancer that has not been discontinued 1 week before start of study treatment.
* Prior adjuvant/neo-adjuvant chemotherapy within 6 months prior to first study treatment. However, if the prior adjuvant/neo-adjuvant chemotherapy was taxane based, patients are excluded if they received their last chemotherapy within12 months prior to first study treatment.
* Prior radiotherapy covering more than 30% of marrow-bearing bone.
* Patients that have received recent radiation therapy that are not recovered from any significant (Grade ≥ 3) acute toxicity prior to study treatment.
* Prior therapy with bevacizumab, sorafenib, sunitinib, or other VEGF pathway-targeted therapy.
* Chronic daily treatment with aspirin
* Chronic daily treatment with corticosteroids, with the exception of inhaled steroids.
* Current or recent treatment with another investigational drug or participation in another investigational study.
* Inadequate bone marrow, liver, renal function
* INR > 1.5 or an aPTT > 1.5 x ULN within 7 days prior to first study treatment.
* Known CNS disease, except for treated brain metastases.
* Patients with concurrent active malignancy
* Pregnant or lactating
* Women of childbearing potential not using effective, non-hormonal means of contraception
* Major surgical procedure (including open biopsy) within 28 days prior to the first study treatment
* Core biopsy or other minor surgical procedure, within 7 days prior to day 1.
* Significant vascular disease within 6 months prior to day 1.
* Any previous venous thrombo-embolism > CTC Grade 3.
* History of haemoptysis
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* Uncontrolled hypertension
* Clinically significant (i.e. active) cardiovasculair disease
* LVEF by MUGA or ECHO < 50%.
* History of abdominal fistula, Grade 4 bowel obstruction or GI perforation, intra-abdominal abscess within 6 months of randomization.
* Serious non-healing wound, peptic ulcer or bone fracture.
* Known hypersensitivity to any of the study drugs or excipients.
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* Psychiatric illness, physical examination or laboratory findings that may interfer with protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  PFS is defined as the time from start of treatment to the documented progression that requires the patient to switch to the next treatment line or to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival second line treatment | 1 year
  To compare the PFS of second line treatment of 8 continuous cycles of chemotherapy with liposomal doxorubicin (or capecitabine) with 8 cycles of intermittent (2 times 4 cycles) chemotherapy with liposomal doxorubicin (or capecitabine);
Objective overall response rate | 1 year
  To compare the objective Overall Response Rate (ORR) between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy in first treatment line, combined with bevacizumab, and in second treatment line.
  ORR calculated as the proportion of patients with a best overall response of confirmed Complete Response (CR) and Partial Response (PR).
Duration of objective response | 1 year
  To compare the Duration of Objective Response (DOR) between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy in first treatment line, combined with bevacizumab, and second treatment line; For the intermittent chemotherapy schedule the first DOR and, if applicable, second DOR in the same treatment line will be accumulated DOR calculated as the time from the date of first documented CR or PR to the first documented progression or death due to underlying cancer
Overall survival | 1 year
  To compare Overall Survival (OS) between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy.
  OS calculated as the time from the date of randomization to the date of death due to any cause or the date of last contact
Safety and tolerability. The total number of grade 3 and 4 adverse events will be analyzed. | 1 year
  To compare the Safety between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy The total number of grade 3 and 4 adverse events will be analyzed as a measure of safety and tolerability
Quality of life measures | 1 year
  To compare the Quality of Life (QoL) between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy.
  Changes in the RAND 36 quality of life scale will be measured
Pharmacoeconomics | 1 year
  To compare the Pharmacoeconomics between 8 continuous cycles of chemotherapy with 8 cycles of intermittent (2 times 4 cycles) chemotherapy.
  Direct medical costs will be calculated using a standard cost method.

CONTACTS AND LOCATIONS:
Overall Officials: F.L.G. Erdkamp, PhD, Principal Investigator — Orbis Medical Centre; M.M.E.M. Bos, PhD, Principal Investigator — RdGG
Locations (1):
- BOOG Study Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: www.boogstudycenter.nl — http://www.boogstudycenter.nl